CLINICAL TRIAL: NCT01576380
Title: A Single-arm, Multi-center, Phase II Study to Evaluate Efficacy and Safety of Dovitinib (TKI258) in Adult Patients With Advanced Scirrhous Gastric Carcinoma That Have Progressed After One or Two Prior Systemic Treatments
Brief Title: A Phase II Study to Evaluate Efficacy and Safety of Dovitinib (TKI258) in Advanced Scirrhous Gastric Carcinoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A1201
Record Dates: First submitted 2012-04-02; First posted 2012-04-12 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Adenocarcinoma, Scirrhous; Linitis Plastica; Stomach Neoplasms; Stomach Diseases; Neoplasms by Site; Neoplasms
Keywords: Solid tumors; Advanced scirrhous gastric carcinoma; Gastric Cancer; Second-line or third-line treatment; VEGF; FGFR; Neoplasms; Gastric Neoplasms; Cancer; Carcinoma; Gastric Diseases; Female Genital Diseases; Tumors; Oral Administration; Capsules; TKI258; TKI-258; TKI 258
MeSH Terms: conditions — Adenocarcinoma, Scirrhous; Linitis Plastica; Stomach Neoplasms; Stomach Diseases; Neoplasms by Site; Neoplasms; Carcinoma; Genital Diseases, Female | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TKI258 (Experimental): TKI258 is dosed on a flat scale of 500 mg, to be administered orally on a 5 days on / 2 days off dosing schedule which will be repeated every week.
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258 — TKI258 is dosed on a flat scale of 500 mg, to be administered orally on a 5 days on / 2 days off dosing schedule which will be repeated every week.
  Other Names: Dovitinib

SUMMARY:
This is a prospective, open-label, single-arm, non-randomized, multi-center, phase II proof of concept (PoC) study with a two-stage design and Bayesian interim monitoring to evaluate efficacy and safety of single agent TKI258 in adult patients with scirrhous gastric carcinoma (SGC) that have progressed after one or two prior systemic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced/metastatic scirrhous gastric carcinoma
* Evidence of diffusely infiltrating gastric lesions and/or at least one measurable extra-gastric lesion
* Patients previously treated with one or two systemic lines
* Documented radiological confirmation of disease progression
* ECOG performance status of 0 to 2
* Male and female patients aged 20 years or greater
* Adequate liver, renal, and hematologic function

Exclusion Criteria:

* Patients who received prior treatment with an FGFR inhibitor
* Patients with known brain metastases or who have signs/symptoms attributable to brain metastases and have not been assessed with radiologic imaging to rule out the presence of brain metastases
* Patients with another primary malignancy within 3 years prior to starting study treatment

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
disease control rate (DCR) | up to 8 weeks after the start date of study treatment
  Eight-week DCR is defined as the proportion of patients with best overall response of CR, PR or SD at the end of Week 8 as per local investigator's assessment.

SECONDARY OUTCOMES:
time to progression (TTP) | baseline and every 4 weeks until Week 17 and every 8 weeks after Week 17 until disease progression
  TTP is defined as the time from the start date of study treatment to the date of event defined as the first documented progression or death due to underlying cancer as per local investigator's assessment.
overall response rate (ORR) | baseline and every 4 weeks until Week 17 and every 8 weeks after Week 17 until disease progress
  ORR is defined as the proportion of patients with best overall response of CR or PR as per local investigator's assessment.
progression free survival (PFS) | baseline and every 4 weeks until Week 17 and every 8 weeks after Week 17 until disease progress
  PFS is defined as the time from the start date of study treatment to the date of event defined as the first documented progression or death due to any cause as per local investigator's assessment.
overall survival (OS) | every 8 weeks until death
  OS is defined as the time from the start date of study treatment to the date of death from any cause.
disease control rate (DCR) per independent central review | up to 8 weeks after the start date of study treatment
  Eight-week DCR is as defined above. An independent central review of the radiological data will be performed and the results will be used for secondary supportive analyses.
time to progression (TTP) per independent central review | baseline and every 4 weeks until Week 17 and every 8 weeks after Week 17 until disease progress
  TTP as defined above. An independent central review of the radiological data will be performed and the results will be used for secondary supportive analyses.
Safety and tolerability of TKI258 | more than 30 days after the last date of study treatment
  Safety will be measured in terms of type, frequency and severity of adverse events according to CTCAE v4.03.
Plasma concentrations of TKI258 | Week 1 Day 1 - Day 2: pre-dose (0 hour), 1, 2, 4, 6, 8, and 24 hour (pre-dose). and Week 4 Day 5 - Week 5 Day 1: pre-dose (0 hour), 1, 2, 4, 6, 8, 24, 48, and 72 hour (pre-dose)
  Pharmacokinetics (PK) of TKI258 at each scheduled time point of single dose and steady dose.
overall response rate (ORR) per independent central review | baseline and every 4 weeks until Week 17 and every 8 weeks after Week 17 until disease progress
  ORR as defined above. An independent central review of the radiological data will be performed and the results will be used for secondary supportive analyses.
progression free survival (PFS) per independent central review | baseline and every 4 weeks until Week 17 and every 8 weeks after Week 17 until disease progress
  PFS as defined above. An independent central review of the radiological data will be performed and the results will be used for secondary supportive analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Japan (8):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Sunto-gun, Shizuoka
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Koto, Tokyo